"Be yourself", educational intervention with chatbot to promote self-determined motivation and prevent adolescent pregnancy: pilot trial protocol

#### **ABSTRACT**

Introduction: Adolescent pregnancy and early initiation of sexual activity is a serious global public health problem, every year, around sixteen million adolescents between 15 and 19 years of age give birth, representing 11% of all births globally. **Objective:** To design a protocol of a pilot Randomized Controlled Trial to evaluate the preliminary efficacy of the "Be Yourself" intervention to increase self-determined motivation to prevent pregnancy in adolescents in secondary education. **Methods:** The protocol was developed based on the Protocol Items: ecommendations for Interventional Trials 2013 (SPIRIT2013) Statement, in the City of Monterrey, Nuevo León, Mexico in 2023. **Results:** The protocol outlined the design of the intervention, structured the content of the sessions using a logic model of intervention, and developed manuals for program facilitators and guides for participants. In addition, a website and a chatbot with Artificial Intelligence were developed, and the strategy for the application of the evaluation instruments was established.

**Keywords**: Self-determination; Teenage Pregnancy; Sexual behaviour; Prevention; Randomized controlled trial.

#### INTRODUCTION

Adolescent pregnancy continues to be a serious public health problem globally, affecting millions of young people every year. The World Health Organization (WHO) and the United Nations Population Fund (UNFPA) report that approximately sixteen million adolescents aged 15 to 19 give birth annually, accounting for 11% of all births. In addition, one in twenty adolescents contracts sexually transmitted infections (STIs) and 3.4 million children under 15 years of age live with Human Immunodeficiency Virus (HIV)<sup>1,2,3</sup>. In Mexico, the rate of teenage pregnancies is the highest in the world, with more than 90% of new STIs in young women and a notable difference in the fertility rate between rural (2.8) and urban (2.01) areas, where 31.2% of young people under 18 years of age in rural areas are already mothers. compared to 18.3% in urban areas<sup>4,5,6</sup>.

The literature reports that some reasons for risky sexual behaviors at this stage are ignorance of the use of contraceptive methods and how STIs are transmitted; lack of communication about sexual issues with parents, friends, and partners; lack of confidence in the proper use of condoms; and lack of sexual autonomy7,8. Different authors indicate that these reasons lead adolescents to some high-risk sexual behaviors, such as the early initiation of sexual relations and sexual relations without using a condom, so that at this stage the risk of unwanted pregnancies and STIs increases 1,9.

Secondary sexual education remains essential to improving adolescent sexual health, as most adolescents attend school, and parents support its inclusion in the curriculum. However, many

adolescent pregnancy prevention programs, created decades ago, address only a limited range of risky behaviors. To increase effectiveness, technology has been integrated into these programs, although evaluations have not always demonstrated the specific impact of these technological components. In addition, it has been noted that programmes that rely solely on in-person education may not be in line with young people's current communication preferences<sup>10,11</sup>.

Recent studies have evaluated technological adaptations in sexual and reproductive health programs, finding that access to websites, apps, and text messages may be promising, although more evaluation is required. Systematic reviews and meta-analyses have comprehensively analyzed interventions to reduce risky sexual behaviors in adolescents, highlighting the importance of psychological approaches based on theories such as Social Cognitive Theory, Planned Behavior Theory, Reasoned Action Theory, and Self-Determination Theory. While most reviews have focused on HIV and STI prevention, some have also addressed pregnancy prevention, often integrating both aspects into their approaches 11,12.

Global evidence indicates that psychological interventions can be effective in reducing risky sexual behaviors and preventing unwanted pregnancies. Adolescent sexual and reproductive health is therefore a national priority. In this context, Rodríguez's Self-Determination Model for Sexual Behavior for the Prevention of Pregnancy in Adolescence (MACSPEA)<sup>13</sup> has proven to be useful in explaining and predicting pregnancy prevention behaviors, considering personal factors such as age, the beginning of sexual life and knowledge about prevention, as well as contextual factors such as sexual communication with parents, friends and partner. In addition, the model includes psychological factors such as intrinsic goals, satisfaction and frustration of basic psychological needs, and self-determined motivation<sup>14,15,16</sup>.

For all the above, an educational intervention was developed based on the MACSPEA model, the six steps of Bartholomew's intervention mapping17 and the stages of the Transtheoretical Model of Change (MTTC) proposed by Prochaska and DiClemente18, in addition to a website that uses artificial intelligence (AI) through a chatbot as a delivery method. This intervention is aimed at adolescents aged 12 to 15 years, with the aim of evaluating the preliminary efficacy of the intervention called "Be yourself" to increase self-determined motivation and prevent pregnancies in secondary school adolescents.

#### MATERIAL AND METHODS

# **Studio Design**

A randomized controlled pilot trial protocol has been developed following the guidelines of the Declaration SPIRIT<sup>19</sup> 2013 and CONSORT<sup>20</sup> criteria, which provides a checklist to ensure quality and completeness in the development of protocols. This protocol corresponds to a randomized controlled pilot trial (RCT) with a pretest-posttest design, which will include a control group (CG) and an experimental group (EG) (Table 1).

**Table 1.** Outline of the design of the Pilot RCT

| Participants | | Assigned<br>Group | Measurement | Application | Measurement<br>1 | Measurement 2 |
|---|---|---|---|---|---|---|
| Teens | | GE-1 | Before | Intervention "Be yourself" | → At the end | 3 months |
| 12 to 15 years | _ | GC- 2 | Before | Habitual | At the end | 3 months |

# Population Characteristics and Eligibility Criteria

The target population of the "Be Yourself" program are adolescents between 11 and 15 years old in secondary schools in Santa Catarina, Nuevo León. Eligibility criteria include being enrolled in a public school with access to a computer lab and internet, residing with your parents, and having become sexually active or not. The sample will be of 150 randomly selected participants. Participation will be assessed using a filter questionnaire, and adolescents will be required to register on the program's website throughout the intervention, with the option to withdraw at any time.

# Sample size

To determine the sample size, the nQuery Advisor statistical package will be used. The aim is to have 150 participants, of which 75 will belong to the CG and 75 to the EG, applying a simple random probability sampling. The sample will be calculated with an error level of .05, a power of 90%, a moderate effect size of .3, considering a loss of 20%.

# Design of the Intervention "Be yourself"

The "Be Yourself" educational intervention was designed to prevent sexual risk in high school adolescents through self-determined motivation. Based on MACSPEA, the model of stages of change and competency-based learning uses a website (<a href="https://www.s-t-mismo.com/">https://www.s-t-mismo.com/</a>) and a chatbot for monitoring and activities (Table 2). The intervention consists of three sessions that address the prevention of adolescent pregnancy and the strengthening of skills. It includes hands-on activities,

role-plays, and interactive sessions on contraceptive methods, effective communication, and informed decision-making. To do this, specialized human resources and specific materials are required for its execution. Manuals were designed for the intervention and training of the facilitator, and activity guides for adolescents<sup>21,14-18</sup>.

**Table 2.** Summary of the content of each session and components of the intervention

| Thematic content | | Time | Components of the intervention | |
|---|---|---|---|---|
| | | Pre-test assessment app | 40 min | Access to the "Be Yourself" page |
| | 1. | What is self-determined motivation?:<br>Discovering our dreams | 60 min | Personal factors 1. Sex |
| First Session | 1. | My Body: Anatomy, Physiology, and Sexual Health. | 60 min | <ul><li>2. Age of onset of sexual life</li><li>3. Pregnancy Prevention</li></ul> |
| | 2. | Navigating relationships: preventing unplanned pregnancy in adolescents. | 60 min | Knowledge |
| | 3. | Exploring Goals and Values to Prevent | 60 min | Contextual factors |
| Second Session | 4. | Unintended Pregnancies Be yourself: stop, think and act; Introduction to Troubleshooting | 60 min | Sexual communication with parents |
| | 5. | Role-play: open dialogue about sexuality | 60 min | <ol> <li>Sexual communication with friends</li> <li>Sexual communication with a partner</li> </ol> |
| — uo | 6. | Navigating the Sea of Healthy Choices:<br>Exploring Our Motivation | 60 min | Psychological factors |
| l Sessi | 7. | 1 0 | 60 min | <ol> <li>Intrinsic and extrinsic motivation</li> <li>Satisfaction and frustration:</li> </ol> |
| Thire | 8. | Negotiating Healthy Choices: Preventing Pregnancy and STIs | 60 min | autonomy, relationships and skills |
| Keep Third Session | 9. | | Continued individual | <ul><li>3. Self-determined motivation,</li><li>4. Behavioral Intent and Sexual<br/>Prevention Behavior</li></ul> |
| | | Post-test assessment app | 40 min | Access to the "Be Yourself" page |
| | | Total, hours | 10 hours 20 | minutes more |

# **Description of the control treatment**

For the GC, two theoretical sessions are planned. In the first, an orientation on sexual health for adolescents will be offered through a one-hour PowerPoint presentation. Topics of anatomy, physiology, biological changes in adolescence and contraceptive methods will be addressed, highlighting their appropriate use and the prevention of teenage pregnancy. In the second session, also one hour, sexual health self-care skills will be developed, discussing the importance of self-care, self-respect, and informed decision-making. There will be a Q&A session to address concerns and reflect on how self-care contributes to a healthy and safe sex life.

#### **Control measures**

# Randomization of participants

Participants will be thoroughly selected to represent the EG. Software will perform a simple, blinded randomization, assigning participants to control or experimental groups. Managers will be informed about the "Be Yourself" sessions, the dates and locations of which will be published on the website and communicated verbally. The sessions will be group, with individual activities on the website and through a chatbot.

# Recruitment

Recruitment for the intervention will take place in February 2025, after the authorization of the educational authorities. Adolescents from the educational institution will be openly invited and their suitability will be evaluated according to inclusion criteria. Those selected will be recorded and assigned to control and experimental groups using an ID to ensure data integrity.

With informed consent, participants will access the website and the chatbot for information and registration. After accepting, they will answer filter questions and receive a detailed explanation of the process. Those who do not qualify will receive a transparent explanation.

On the website, participants will record their personal data for effective communication and reminders. They will be informed about the royalties of the program at the end of the project, motivating them to participate in all activities. The information will be stored securely for one year.

# Measurements and data collection

Data collection for the study will include the use of a specifically designed Personal Data Card, which will collect information about the sexuality, marital status, and education of the participants. A variety of scales will be used to measure aspects related to adolescent sexual health and behavior. The Sexual and Reproductive Health Knowledge Scale, Cronbach's alpha between .77 and .81<sup>21</sup>, will assess knowledge in these areas, while the Sexual Issues Communication Instrument, Cronbach's alpha from .89 to .95, will analyze sexual communication between parents, friends, and partners<sup>22</sup>. The Aspirations Index, alpha greater than .78 and .94, will measure life goals, and the Basic Psychological Needs Satisfaction and Frustration Scale will have alphas of .90 and .86<sup>23</sup>.

The Behavior Regulation Questionnaire, adapted to the Mexican context, will assess behavior regulation to prevent pregnancy, with alphas between .66 and .93<sup>24</sup>. Likewise, the Sexual Activity Intention Scale and the Sexual Activity Scale will assess sexual intentions and behaviors, respectively, with alphas from .83 to .88 and .74 to .86<sup>25</sup>. The Sexual and Reproductive Health

Practices Scale, which examines pregnancy prevention behavior, with alphas of .92, .77, .81 and .87 in its different adaptations<sup>26</sup>.

The "Scale for the Assessment of Change on Sexual Behavior in Adolescents" 27 will be adapted and validated, ensuring its reliability. To assess the acceptability and feasibility of the "Be Yourself" intervention, aspects such as participant satisfaction, meeting expectations, and facilitator quality will be analyzed, along with participant recruitment, screening, randomization, and retention procedures.

# Participant Retention Plan and Follow-Up

The retention plan for the "Be yourself" intervention includes the delivery of T-shirts and caps with the logo of the program at the end, weekly sessions to avoid information saturation and a three-month follow-up. Data collection will be done through the website using digital tools to assess the effectiveness and acceptability of the program. The fidelity of the intervention will be ensured by training the principal investigator in self-determination theory and developing supporting manuals and guides. Figure 1 presents diagram CONSORT<sup>20</sup>, which details the eligibility criteria, intervention, and evaluation of sessions before, after, and during follow-up at three months.

Figure 1. CONSORT diagram of the "Be yourself" intervention



This study complies with the ethical regulations of the Regulations of the General Health Law, ensuring respect for the dignity and rights of the participants. The protocol has been approved by the Ethics and Research Committee of the Faculty of Nursing of the Autonomous University of Nuevo León, with registration number FAEN-D-2021. Informed consent will be obtained from the parents and assent from the adolescents. Participation will be explained in detail to parents and teens, including risks and benefits. The research will be suspended if there is a risk to the health of the participants or if they wish to withdraw <sup>28</sup>.

# Data analysis plan

The research will use statistical software SPSS version 26.0 for data processing. The analysis will begin with the Kolmogorov-Smirnov test to evaluate the distribution of the data and determine the suitability of applying parametric or nonparametric tests. The statistical analysis will include a descriptive level, using percentages, means, and standard deviation, to assess feasibility and acceptability. For hypotheses, inferential tests such as paired sample t-test, ANOVA, and Mann-Whitney U will be used to examine knowledge about pregnancy prevention, sexual communication, motivation, satisfaction of psychological needs, sexual intention, pregnancy prevention behavior, and stages of change in sexual behavior<sup>29</sup>.

Table 3 describes the objectives and hypotheses proposed in this study, both descriptive and inferential statistics will be used

**Table 3**. Statistical analysis by objective and/or hypothesis

| Objective | Analysis | Statistical |
|---|---|---|
| 1 Examining feasibility | Descriptive | Measures of frequency, central tendency, and dispersion: percentages, means, ranges, Standard Deviation, confidence intervals, recruitment and retention rates. |
| 2 Analyze acceptability | Descriptive | Percentages, means, ranges, Standard<br>Deviation, confidence intervals,<br>recruitment and retention rates |
| Hypothesis | Analysis | Statistical |
| <ul> <li>3 Hypothesized results:</li> <li>H 1. Knowledge about Pregnancy Prevention</li> <li>H 2. Sexual Communication Parent, Friends &amp; Partner.</li> <li>H 3. Intrinsic and extrinsic motivation</li> <li>H 4. Satisfactory and Frustration of NPBs (autonomy, relationship and competencies)</li> <li>H 5. Self-Determined Motivation</li> <li>H 6. Intention in Sexual Activity</li> <li>H 7. Pregnancy Prevention Sexual Behavior</li> <li>H 8. Stages of Change for Sexual Behavior</li> </ul> | Inferential | t-test of paired or ANOVA samples<br>Test de Friedman<br>Test de Wilcoxon<br>U de Mann-Whitney |

#### EXPECTED RESULTS

The protocol of the "Be Yourself" intervention includes the structural design of the sessions, the development of two facilitator manuals and a participant workbook, and the creation of a web page with a chatbot based on OpenAI's GPT. The intervention is expected to increase adolescents' self-determination to abstain from sexual activity, improve their positive attitude toward sexuality, and expand their knowledge about pregnancy prevention. In addition, a greater adoption of preventive behaviors is anticipated compared to those who do not participate, which would suggest a positive impact on sexual decision-making.

#### FINANCING

This project did not receive any funding

# **DECLARATION OF CONFLICTS OF INTEREST**

The author declares that they have no conflict of interest

# **REFERENCES**

- World Health Organization (WHO)/PAHO. Syndromic management of sexually transmitted infections. 2022. ISBN 9789243593401. [Accessed July 19, 2024]. Available in: <a href="https://www.paho.org/es/temas/infecciones-transmision-sexual/manejo-sindromico-infecciones-transmision-sexual">https://www.paho.org/es/temas/infecciones-transmision-sexual/manejo-sindromico-infecciones-transmision-sexual</a>
  - UNFPA. Systematization of scientific evidence on Comprehensive Sexuality Education.
     Updated version with new evidence about out-of-school HIE. UNFPA Regional Office for Latin America and the Caribbean, Panama. 2020. [Accessed July 19, 2024]. Available in: <a href="https://www.aprofaeduca.cl/wp-content/uploads/2021/08/Sistematizacio%CC%81n-de-evidencias-cienti%CC%81ficas-sobre-la-Educacio%CC%81n-Integral-de-la-Sexualidad.pdf">https://www.aprofaeduca.cl/wp-content/uploads/2021/08/Sistematizacio%CC%81n-de-evidencias-cienti%CC%81ficas-sobre-la-Educacio%CC%81n-Integral-de-la-Sexualidad.pdf</a>
- 1. The United Nations Population Fund (UNFPA) and the United Nations Population Fund (UNFPA) are promoting a pilot project for the prevention of teenage pregnancies in the Xochimilco Mayor's Office in Mexico City. 2022. UNFPA Mexico. [Accessed July 19, 2024]. Available in: <a href="https://mexico.unfpa.org/es">https://mexico.unfpa.org/es</a>
- 1. Mungai Gakuo A. Factors influencing the occurrence of adolescent pregnancies among adolescent girls attending the antenatal clinic at Kiambu Health Centre in Kenya [Master's thesis]. International University of Health Sciences. 2023. Available in:

  <a href="http://dspace.ciu.ac.ug/handle/123456789/265?show=full">http://dspace.ciu.ac.ug/handle/123456789/265?show=full</a>
  - 2. Xie Y, Wang X, Mu Y. Characteristics and adverse outcomes of Chinese adolescent pregnancies between 2012 and 2019. Sci Rep. 2021; 11:12508. Disponible en:

# https://doi.org/10.1038/s41598-021-92037-x

- 3. Logie CH, Lys CL, Fujioka J, MacNeill N, Mackay K, Yasseen III AS. Sexual practices and condom use among a sample of Northern and Indigenous adolescents in Northern Canada: cross-sectional survey results. BMJ Sex Reprod Health. 2020;45(2):147-154. Disponible en: <a href="https://doi.org/10.1136/bmjsrh-2018-200174">https://doi.org/10.1136/bmjsrh-2018-200174</a>
- Logie CH, Lys CL, Mackay K, MacNeill N, Pauchulo A, Yasseen AS. Syndemic factors associated with safer sex efficacy among Northern and Indigenous adolescents in Arctic Canada. Int J Behav Med. 2021;26(4):449-453. Disponible en:
   <a href="https://doi.org/10.1007/s12529-019-09797-0">https://doi.org/10.1007/s12529-019-09797-0</a>
- Molina AM, Gómez RA, Díaz CE, Soto MA. Condicionantes y consecuencias sociales del embarazo en la adolescencia. 2019;45(2):1-21. Disponible en: http://scielo.sld.cu/pdf/gin/v45n2/1561-3062-gin-45-02-e218.pdf
- 6. Coyle K, Anderson PM, Laris BA, Barrett M, Unti T, Baumler E. A group randomized trial evaluating High School FLASH, a comprehensive sexual health curriculum. J Adolesc Health [Internet]. 2021 Apr 1;68(4):686-695. Disponible en: <a href="https://doi.org/10.1016/j.jadohealth.2020.12.005">https://doi.org/10.1016/j.jadohealth.2020.12.005</a>
- 7. Manlove J, Cook E, Whitfield B, Johnson M, Martínez-García G, Garrido M. Short-term impacts of Pulse: an app-based teen pregnancy prevention program for Black and Latinx women. J Adolesc Health [Internet]. 2020;66(2):224-232. Disponible en: https://doi.org/10.1016/j.jadohealth.2019.08.017
- 8. Swain LT, Malouff JM, Meynadier J, Schutte NS. Psychological interventions decrease unintended pregnancies: a meta-analysis of randomized controlled trials. Br J Health Psychol [Internet]. 2023;28(2):567-585. Disponible en: https://doi.org/10.1111/bjhp.12641
- 9. Marseille E, Mirzazadeh A, Biggs MA, Miller AP, Horváth H, Lightfoot M, et al. Effectiveness of school-based teen pregnancy prevention programs in the USA: a systematic review and meta-analysis. Prev Sci [Internet]. 2018;19(4):468-489. Disponible en: https://doi.org/10.1007/s11121-017-0861-6
- 10. Rodríguez Vázquez N. Modelo de autodeterminación para la conducta sexual de prevención del embarazo en la adolescencia [Tesis doctoral]. Universidad Autónoma de Nuevo León. 2021. Disponible en: <a href="http://eprints.uanl.mx/22154/">http://eprints.uanl.mx/22154/</a>
- 11. Ryan RM, Deci EL. Self-Determination Theory: Basic Psychological Needs in Motivation,

- Development, and Wellness. Guilford Publications; 2018.
- 12. Rotta I, Rodríguez AT, Fernández BD, De Mendoza Lima T. Effectiveness of strategies to delay sexual activity onset to prevent pregnancy in the adolescence: a... ResearchGate [Internet]. 2023 [consultado el 19 de julio de 2024]. Disponible en: <a href="https://www.researchgate.net/publication/370119693">https://www.researchgate.net/publication/370119693</a> Effectiveness of strategies to dela y sexual activity onset to prevent pregnancy in the adolescence a systematic revie w
- Garzón-Orjuela N, Samacá-Samacá D, Moreno-Chaparro J, Ballesteros-Cabrera M, Eslava-Schmalbach J. Effectiveness of sex education interventions in adolescents: an overview. Compr Child Adolesc Nurs. 2020;44(1):15-48.
   <a href="https://doi.org/10.1080/24694193.2020.1713251">https://doi.org/10.1080/24694193.2020.1713251</a>
- 14. Bartholomew LK, Parcel GS, Kok G, Gottlieb NH, Fernández ME. Planning Health Promotion Programs: An intervention mapping approach. 4th ed. San Francisco: Jossey-Bass; 2016.
- 15. Prochaska JO, DiClemente CC, Norcross JC. In search of how people change: applications to addictive behaviors. Addict Nurs Netw. 1992;5(1):2-16.
- 16. Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gøtzsche PC, Krleža-Jerić K, et al. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013;158(3):200-207.
- 17. Thabane L, Hopewell S, Lancaster GA, Bond CM, Coleman CL, Campbell MJ, et al. Methods and processes for development of a CONSORT extension for reporting pilot randomized controlled trials. Pilot Feasibility Stud. 2016;2:25. PMID: 27965844.
- 18. Vargas Ruiz R. Conocimientos, actitudes y prácticas en salud sexual y salud reproductiva: propuesta de una escala psicométrica. Instituto de Estudios Sociales en Población (IDESPO); 2013.
- 19. Hutchinson MK, Cooney TM. Patterns of parent-teen sexual risk communication: implications for intervention. Fam Relat. 1998;47(2):185-194.
- 20. Del Valle M, Matos L, Díaz A, Pérez MV, Vergara J. Propiedades psicométricas de la Escala de Satisfacción y Frustración de Necesidades Psicológicas (ESFNPB) en universitarios chilenos. Propós Represent. 2018;6(1):301-350.
- 21. González-Cutre D, Sicilia A, Fernández A. Hacia una mayor comprensión de la motivación en el ejercicio físico: medición de la regulación integrada en el contexto español.

- Psicothema. 2010; 22:841-847.
- 22. Bello-Villanueva AM, Palacio J, Rodríguez-Díaz M, Oviedo-Trespalacios O. Medición de la intención en la actividad sexual en adolescentes: una aproximación de acuerdo al género del Caribe colombiano. Terap Psicol. 2013;31(3):343-353. <a href="https://dx.doi.org/10.4067/S0718-48082013000300009">https://dx.doi.org/10.4067/S0718-48082013000300009</a>
- 23. Vargas E, Trujillo Barrera V. Escala de actividad sexual: un instrumento para predecir el inicio temprano de relaciones sexuales. Behav Psychol/Psicologia Conductual. 2002;18(3):591+. Disponible en:

  <a href="https://link.gale.com/apps/doc/A314254342/AONE?u=anon~565fae67&sid=googleScholar&xid=1cb58c1b">https://link.gale.com/apps/doc/A314254342/AONE?u=anon~565fae67&sid=googleScholar&xid=1cb58c1b</a>
- 24. Cabrera AG. El modelo transteórico de comportamiento en salud. Rev Fac Nac Salud Pública. 2000;18(2):129-138.
- 25. Secretaría de Salud [SSA]. Reglamento de la Ley General de Salud en Materia de Investigación para la Salud, México. Ciudad de México: SSA; 2014.
- 26. Merrill KG, Atujuna M, Emerson E, Blachman-Demner D, Bray BC, Bekker LG, et al. Preliminary effectiveness and implementation outcomes of the IMARA-South Africa sexual health intervention on adolescent girls and young women: a pilot randomized trial. PLOS Glob Public Health [Internet]. 2023 Feb 15;3(2). Disponible en: <a href="https://doi.org/10.1371/journal.pgph.0001092">https://doi.org/10.1371/journal.pgph.0001092</a>
- 27. Purcell C, McDaid L, Forsyth R, Simpson SA, Elliott L, Bailey JV, et al. A peer-led, school-based social network intervention for young people in the UK, promoting sexual health via social media and conversations with friends: intervention development and optimisation of STASH. BMC Public Health [Internet]. 2023 Apr 11;23(1). Disponible en: <a href="https://doi.org/10.1186/s12889-023-15541-x">https://doi.org/10.1186/s12889-023-15541-x</a>
- 28. Roman Lay AA, Fujimori E, Simões Duarte L, Vilela Borges AL. Prevalence and correlates of early sexual initiation among Brazilian adolescents. PLoS One. 2021;16(12). <a href="https://doi.org/10.1371/journal.pone.0260815">https://doi.org/10.1371/journal.pone.0260815</a>
- 29. IBM Corp. IBM SPSS Statistics for Windows, Versión 22.0. [Software de computación]. Armonk, NY: IBM Corp; 2013.

# Logical Model of the "Be Yourself" Intervention

#### **Problem**

Self-determined motivation for adolescent pregnancy prevention.

Meta

That adolescents achieve the stage of action and maintenance of self-determined motivation to prevent adolescent pregnancy.

# Justificatio n

Situation-Specific Theory of Self-Determined Motivation for the Prevention of Pregnancy, Transtheoretical Model of Change (Prochaska and Di Clemente) and the Competency-Based Learning Model (Herreras, 1970)

#### Assumptions

- a. Adolescents in the precontemplation stage may not recognize themselves at risk for pregnancy if they lack awareness of the associated consequences and risks.
- If teens don't have enough knowledge about pregnancy prevention, condom use, and birth control, they're likely to stay in the contemplation stage.
- c. A lack of self-determined motivation toward abstinence and condom use can hinder adolescents' transition to the preparation stage.
- d. A lack of sexual communication with parents, friends, and partners can make it difficult for teens to move into the action stage, where they are expected to implement changes in sexual behavior and behavior.
- e. Lack of sexual autonomy, inability to negotiate condom use, and abstinence may be factors influencing adolescents' ability to **sustain** positive changes in sexual behavior and behavior.
- f. Adolescents are more likely to change their sexual behavior and behavior if the intervention and prevention messages are personalized, affectionate and supportive.
- Maintaining an effective self-determined motivation based on learning is essential

## Human: Researcher. research assistant Financial: Operating budget for the production of the material. **Space:** Computer room of the educational institution Materials: didactic and recreational materials for the intervention. Access to the web platform Interactive digital educational material. Technical support to

solve possible

problems.

Entrance

Resources

# to

#### Activities Outputs **Session 1:** Getting to know 1. "Be Yourself" yourself, steps to achieve faithfully your "Be Yourself" goals implemented. Knowledge and awareness 2. Videos viewed on 1. What is Self-Determined web platform Motivation?: Discovering 3. Participants Our Dreams discuss condom 2.My Body: Anatomy, use and Physiology and Sexual negotiation Health. 4. There is a Problem solving, discussion about negotiation. abstinence and 3. Navigating Relationships: prevention of Preventing Unwanted Teen pregnancy Pregnancy. 5. Negotiation and **Session 2:** Building Personal rejection skills Commitments: Conduct, are practiced Behavior, and Sexual through role Communication plays. 1. Exploring Goals and 6. Acquired Values to Prevent problem skills. Unintended Pregnancies 7. Self-confidence 2. Be yourself: stop, think in decisionand act; Introduction to making Troubleshooting Practice sexual 3. Role-Play: Open Dialogue communication on Sexuality **Session 3:** Empowerment and Concrete Actions:

**Outputs** 

#### Results

#### Primary

- 1. Increase in Self-Determined Motivation Indices to Prevent Adolescent Pregnancy (H5).
- 2.Increased Level of Knowledge about Pregnancy Prevention (H1).
- 3.Improved Communication on Sexual Issues (H2.
- 4. Change in Life Goals (H3): Significant increase in orientation toward intrinsic life goals (such as personal and academic development).
- 5. Satisfaction of Basic Psychological Needs: autonomy, relationships and competence. (H4).

#### Secondarys

- 1. Intention to Risk and Protect (H6):
  Significant decrease in intention to risk
  (such as willingness to have
  unprotected sex) and significant
  increase in intention to protect (such as
  use of contraception and protection
  against STIs).
- 2.Frequency of Nonsexual Sexual and Affection Behaviors (H7): Significant decrease in the frequency of risky sexual behaviors and increase in the frequency of nonsexual affection

| for the consolidation of change in the sexual conduct and behavior of adolescents. h. Believing in themselves and their abilities, feeling valued, and having opportunities to practice skills with the support of parents, friends, and partners are key factors in preventing relapses of risky sexual behaviors and behaviors. | improving negotiation and rejection skills 1. Navigating the Sea of Healthy Choices: Exploring Our Motivation. 2. My space, my decisions exploring our needs. 3. Negotiating Healthy Choices: Preventing | behaviors (such as holding hands and kissing on the mouth). 3. Highly preventive behavior with favorable attitudes and behaviors toward pregnancy prevention (H8) 1. Intention and Willingness to Change Sexual Behavior in the Next Three Months (H9) |
|---|---|---|
| | Pregnancy and STIs | |

#### **Products**

Session 1: Getting to know yourself, steps to achieve your "Be Yourself" goals (Knowledge and awareness)

- 1. The adolescent becomes aware of pregnancy prevention and what is involved in increased knowledge of the risks associated with sexual activity, as well as an understanding of the importance of family planning and the prevention of unintended pregnancy.
- 2. Detailed knowledge about the correct use of condoms and awareness of their importance in protecting against STIs are key results in promoting sexual health.
- 3. Improved negotiation skills are reflected in an increased ability to communicate and reach agreements, accompanied by the development of empathic skills and a broader understanding of others' perspectives.

Session 2: Building Personal Commitments: Conduct, Behavior, and Sexual Communication

- 1. Exploring Goals and Values: Teens identify personal goals and strategies to prevent pregnancy through hands-on exercises and role-playing.
- 2. Problem-solving: Communication skills and informed decision-making are developed in relationships, focusing on values and limits.
- 3. Role play: Open communication about sexuality is practiced with parents, friends and partners, evaluating progress and challenges.

Session 3: Empowerment and Concrete Actions: improving negotiation and rejection skills

- 1. Teens will create a "Negotiation and Rejection Skills Guide." This guide would include specific strategies learned during the session, practical tips for coping with challenging situations in preventing unintended pregnancy.
- 2. Adolescents participate in the "Motivational Campaign on Sexual Health", promoting the importance of personal empowerment, informed decision-making and self-motivation on issues related to sexual health. This campaign could include inspirational messages, testimonials, and helpful resources to foster self-determination among peers.
- 3. "Interactive Simulation with Chatbot", which simulates situations of negotiation and rejection in the context of sexual relations and prevention of unplanned pregnancy, allows adolescents to practice and reinforce the skills learned, providing instant feedback on their choices and decisions.